CLINICAL TRIAL: NCT00516282
Title: A Phase I/II Trial of Cloretazine® (VNP40101M) and Temodar® (Temozolomide) for Patients With Malignant Glioma in First Relapse or Progression
Brief Title: VNP40101M and Temozolomide in Treating Patients With Progressive or Relapsed Malignant Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The pharmaceutical collaborator filed for bankruptcy and as a result, the study was unable to move into the phase II portion.
Sponsor: Northwestern University (Other)
Collaborators: Vion Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 07C1
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Glioma | interventions — laromustine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CLORETAZINE — CLORETAZINE will be administered intravenously on day 7. The starting dose of CLORETAZINE will be 100 mg/m2 given within 3 hours after the last dose of Temodar on day 7. CLORETAZINE will be given as an IV infusion over 15-30 minutes via a freely flowing peripheral or central intravenous line. CLORETAZINE will be escalated by 50 mg/m2 for the second cohort then by 25 mg/m2 increments in the following cohorts of 3-6 patients using a standard phase I trial design until a MTD is determined. If dose level 2 has two DLTs then patients will be accrued to a new dose level of 125 mg/m2. Prior to receiving Cloretazine, blood will be drawn for gene methylation studies.
  Other Names: VNP40101M
Drug: temozolomide — Temozolomide will be given orally at a dose of 75mg/m2 daily on day 1 through 7. There will be no dose modification for this agent. Prior to receiving Temozolomide, blood will be drawn for gene methylation studies.
  Other Names: Temodar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide and VNP40101M, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Temozolomide may also stop the growth of tumor cells by blocking blood flow to the tumor.

PURPOSE: This phase I/II trial is studying the side effects and best dose of VNP40101M when given together with temozolomide and to see how well it works in treating patients with progressive or relapsed malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose (MTD) of VNP40101M when administered with temozolomide in patients with progressive or relapsed (first relapse) malignant glioma. (Phase I)
* To record the toxicities of VNP40101M when administered with temozolomide. (Phase I and II)
* To measure the level of AGT expression in peripheral blood monocytes before treatment with temozolomide and just prior to the administration of VNP40101M. (Phase I and II)
* To determine MGMT methylation status as well as other methylation patterns in blood and tissue from patients treated with this regimen and correlate with outcome. (Phase I and II)
* To determine the 6- and 12-month progression-free survival rates of patients treated with this regimen. (Phase II)
* To determine overall survival of patients treated with this regimen. (Phase II)
* To determine the complete and partial response rates in patients treated with this regimen. (Phase II)
* To determine CSF penetration of VNP40101M once the MTD is reached from phase I and correlate with serum/plasma pharmacokinetics. (Phase II)

OUTLINE:

* Phase I: Patients receive oral temozolomide on days 1-7 and VNP40101M IV over 15-30 minutes 2 hours after the last dose of temozolomide on day 7. Treatment repeats every 7 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of VNP40101M until the maximum tolerated dose (MTD) is determined The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

* Phase II: Patients receive oral temozolomide and VNP40101M as in phase I. VNP40101M is given at the MTD determined in phase I.

In both phases, patients complete the Functional Assessment of Cancer Therapy-Brain (FACT-BR) questionnaire on day 1 of each course.

Blood is collected for in vitro isolation of mononuclear cells for analysis of O^6 alkylguanine DNA alkyltransferase on days 1 and 7 of course 1. Blood, plasma, CSF, and formalin-fixed paraffin-embedded tissue blocks are collected for gene methylation studies, including MGMT, at baseline and on day 1 of each course.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically proven malignant glioma including any of the following:

  * Glioblastoma multiforme
  * Gliosarcoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant astrocytoma not otherwise specified
* Unequivocal evidence of tumor recurrence or progression by MRI or CT scan with contrast
* No more than one relapse
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  * More than 2 weeks from surgery and have recovered from the effects of surgery
  * Evaluable or measurable disease following resection of recurrent tumor is not mandated for eligibility into the study if a treatment failure can be evaluated
  * Enhanced CT scan/ MRI should be done no later than 96 hours in the immediate post-operative period or 4-6 weeks post-operatively

    * If the 96-hour scan is more than 2 weeks from registration, the scan needs to be repeated
    * A baseline scan should be performed within 14 days prior to registration and on a steroid dosage that has been stable for 5 or more days otherwise a new baseline MRI/CT is required
    * The same type of scan (i.e., MRI or CT scan) must be used throughout the period of protocol treatment for tumor measurement
* Must have failed prior external-beam radiotherapy
* Must have failed one prior systemic treatment with chemotherapy or biologic agents

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status 60-100%
* Life expectancy > 12 weeks
* WBC > 3,000/mm³
* ANC > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 10 mg/dL
* AST and ALT < 4 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* Creatinine < 1.5 times ULN
* Fertile patients must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device)
* Negative pregnancy test
* Not pregnant or nursing

Exclusion criteria:

* Active uncontrolled bleeding
* Active infection of any kind
* Unwilling or unable to follow protocol requirements or to give informed consent
* Active heart disease including any of the following:

  * Myocardial infarction within the past 3 months
  * Uncontrolled arrhythmias
  * Uncontrolled coronary artery disease
  * Uncontrolled congestive heart failure
* Known HIV-positive patients (HIV testing is not required)
* History of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) unless in complete remission and off all therapy for that disease for a minimum of 3 years

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* Recovered from prior therapy
* At least 2 weeks since prior vincristine
* More than 4 weeks since prior cytotoxic therapy (6 weeks for nitrosoureas)
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior experimental biologic agents (e.g., EGFR inhibitors, etc)
* More than 3 weeks since prior procarbazine administration
* More than 2 weeks since prior non-cytotoxic agents (e.g., interferon, tamoxifen, thalidomide, or isotretinoin)

  * Radiosensitizer does not count
* At least 2 weeks since prior and no concurrent enzyme inducing anticonvulsants

  * If patient is on an enzyme inducing anticonvulsant, they may be converted to a non-enzyme inducing anticonvulsant

Exclusion criteria:

* Any other concurrent standard or investigational treatment for cancer, or any other investigational agent for any indication
* Concurrent disulfiram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
MTD of CLORETAZINE | At the end of phase one
  To determine the MTD of CLORETAZINE when administered with Temodar® in patients with malignant gliomas in first or second relapse
Progression-free survival rate | End of Phase II
  To determine the 6 and 12 month progression-free survival rate.

SECONDARY OUTCOMES:
Toxicities of CLORETAZINE when administered with Temodar®. | Adverse events are monitored at screening/baseline;day one; termination visit; followup until death.
  To record the toxicities of CLORETAZINE when administered with Temodar®.
  (Toxicity is assessed continuously through routine medical monitoring of the patient throughout each cycle and all adverse events are recorded cumulatively on the case report forms).
MGMT Methylation Status | Baseline and day seven of every cycle
  To determine MGMT methylation status as well as other methylation patterns in blood correlate with outcome.
Determine overall survival | All patients will be followed until death
  To determine overall survival.
Response rate to CLORETAZINE after Temodar® in patients with malignant gliomas in first or second relapse | Day one of every cycle
  To determine the response rate to CLORETAZINE after Temodar® in patients with malignant gliomas in first or second relapse.
Record the toxicities of CLORETAZINE when administered after Temodar | Continuously after the first dose;within thirty days of each administration of investigational agent
  To record the toxicities of CLORETAZINE when administered after Temodar®
Measure the level of AGT expression | Day seven of every cycle
  To measure the level of AGT expression in peripheral blood monocytes before treatment with Temodar® and just prior to the administration of CLORETAZINE.
CSF penetration of CLORETAZINE | Day seven of cycle one of Phase 2 only
  To determine CSF penetration of CLORETAZINE once the MTD is reached from phase I and correlate with serum/plasma PK

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Raizer, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Northwestern University, Chicago, Illinois